CLINICAL TRIAL: NCT05077592
Title: Addition of Pre-wound Closure Povidone Iodine Wash Versus Direct Wound Closure Effect on Surgical Site Infections: A Randomized Controlled Trial
Brief Title: Addition of Pre-wound Closure Povidone Iodine Wash Versus Direct Wound Closure Effect on Surgical Site Infections
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Walid Ahmed Abdel-Ghany, Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: POV-2021
Record Dates: First submitted 2021-09-19; First posted 2021-10-14 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Surgical Site Infection; Surgical Wound Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Povidone-Iodine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: A statistician not directly involved in the study or analysis will prepare a computer-generated randomization sequence. No blocking will be used. The sequence will be provided to the trialists in the form of serially numbered opaque envelopes containing details of either the intervention or the control and a random identifier.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Direct Wound closure
- Intervention (Active Comparator): The use of 10% surgical povidone iodine to wash the wound directly after fascial closure and before wound closure
  Interventions: Drug: 10% Povidone Iodine

INTERVENTIONS:
Drug: 10% Povidone Iodine — Povidone-iodine is a topical antiseptic agent used for the treatment and prevention of infection in wounds.
  Other Names: betadine
  Arms: Intervention

SUMMARY:
A Randomized controlled trail to To assess the efficacy of povidone-iodine wash before wound closure in preventing surgical site infections.

DETAILED DESCRIPTION:
Surgical site infections are post-operative infections of the incision or organ or space that was included in the surgical field. Incisional surgical site infections (SSIs) are a growing healthcare challenge.

Currently, up to 10% of surgical procedures may be complicated by an SSI [3]. Not only do SSIs lead to worse patient outcomes, but they also account for a large proportion of healthcare expenditure.

In the United Kingdom alone, SSIs are estimated to cost the National Health Service 1 billion pounds annually.

The problem is further compounded in low- and middle-income countries (LMICs) where the prevalence of antibiotic-resistant infections is increasing, and national healthcare budgets are strained.

In fact, SSIs are estimated to account for additional costs of up to $30,000 in LMICs.

The global crisis of drug-resistant bacteria has further highlighted the need for more effective perioperative preventive strategies to minimize healthcare-associated resistant infections.

Optimal surgical antisepsis is critical in reducing the incidence of SSIs, and therefore in reducing the use of postoperative antibiotics.

Recently, there has been a renewed interest in using povidone-iodine (PVI) intraoperative wound irrigation to achieve this goal. The choice of PVI is especially suitable for LMICs where the availability of chlorhexidine preparations may be limited by scarce resources.

A possible adjunctive role of pre-wound closure PVI irrigation in reducing incisional SSIs is still unclear.

A meta-analysis by López-Cano et al. analyzed data of 7,601 patients and found a reduction in overall SSI rate. However, the heterogeneity and uncertain quality of most studies limited the synthesis of conclusive evidence.

The possible benefits of irrigating the surface of an open incision include local antimicrobial effect, physical removal of debris and dilution of contamination. Recent guidelines have all emphasized the lack of sufficient evidence on intraoperative use of PVI.

The investigators aim to conduct a randomized controlled trial in Ain Shams University Hospitals to compare the effect of adding PVI wash prior to skin closure to direct wound closure on reducing the rates of SSIs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years old)
* Open and minimally invasive surgeries
* Emergency (any unplanned admission) and elective (planned admission) surgical procedures
* Clean, Clean-Contaminated, Contaminated, Dirty wounds
* Inclusion surgery list according to Current Procedural Terminology (CPT) National Healthcare Safety Network (NHSN) operative procedure code mapping

Exclusion Criteria:

* Povidone-iodine allergy
* Surgeries for infected wounds.
* Exclusion surgery list according to Current Procedural Terminology (CPT) National Healthcare Safety Network (NHSN) operative procedure code mapping.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 760 (Estimated)
Dates: Start 2021-09-18 (Actual); Primary Completion 2021-12-18 (Estimated); Study Completion 2022-01-18 (Estimated)

PRIMARY OUTCOMES:
Surgical Site Infection Incidence | 30 days
  Using the CDC Checklist for Superficial and deep Surgical site infection.

SECONDARY OUTCOMES:
Post-operative morbidity and mortality | 30 Days
  Using the Clavien-Dindo classification system
Length of hospital stay | 30 Days
  in days using the hospital records
Readmission and reoperations related to Surgical site infection | 30 Days
  Using the hospital records, Number of reoperations and readmissions due to surgical site infection.
Infectious complications | 30 Days
  Using qSOFA and SOFA score. such as Sepsis, septic shock, multiple-organ dysfunction syndrome, wound dehiscence
Microbiology culture and sensitivity results | 30 Days
  A microbiology report that contains the exact pathogen strain and antibiotic sensitivity report.
Local adverse events for povidone-iodine application | 30 Days
  Symptoms and sings
Cost analysis | 30 Days
  In terms of extra hospital stay days and readmission days costs.

CONTACTS AND LOCATIONS:
Overall Officials: Waleed AbdelGhany, Professor, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2021-09-11): https://cdn.clinicaltrials.gov/large-docs/92/NCT05077592/Prot_000.pdf
  • Informed Consent Form (2021-06-13): https://cdn.clinicaltrials.gov/large-docs/92/NCT05077592/ICF_001.pdf